CLINICAL TRIAL: NCT01988129
Title: Fire Fighter Fatigue Management Program: Operation Healthy Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Federal Emergency Management Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Andrew Czeisler, MD, PhD, Charles A Czeisler, Ph.D., M.D.,, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-000697
Record Dates: First submitted 2010-07-27; First posted 2013-11-20 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Shift-Work Sleep Disorder; Insomnia; Restless Leg Syndrome; Obstructive Sleep Apnea; Impaired Driving; Injuries
Keywords: sleep; firefighter; fire; apnea; insomnia; shift; narcolepsy; restless leg; rls; fatigue; actigraph; actigraphy; actiwatch; safety; sleepiness; sleepy; work; hours; Federal Emergency Management Agency; drowsy
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Restless Legs Syndrome; Sleep Apnea, Obstructive; Wounds and Injuries; Apnea; Narcolepsy; Fatigue; Sleepiness | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Workplace-based fatigue risk management program consisting of sleep health education and sleep disorders screening. The 32 fire department stations were paired according to the previous calendar years' workload. One station from each pair was randomly assigned to receive the intervention program. Sleep education sessions were scheduled according to station. On the education day(s) assigned to that stations, all personnel present that day were instructed to attend, and 542/601 did so.
  Interventions: Other: Sleep disorders education and screening
- Control (No Intervention): Current practice. Firefighters in the Control Stations continued their normal role and were not invited to attend the sleep education and sleep disorders screening program. There was no formal contact with the control group.
  As part of normal operational requirements, a small number of firefighters are reassigned to other stations each day and therefore 18/588 firefighters from control stations happened to be reassigned to an intervention station on the day of the education session and attended the session.

INTERVENTIONS:
Other: Sleep disorders education and screening — Firefighters were instructed to attend an education presentation as operations allowed which provided information on firefighter mortality, fatigue-related health hazards and discussed the importance of sleep, and also included strategies to improve sleep hygiene and how to use caffeine and naps effectively to promote alertness. Firefighters were then invited to complete a voluntary sleep disorders screening survey. This survey used validated, self-report screening tools for obstructive sleep apnea, moderate to severe insomnia, restless legs syndrome and shift work disorder. All of those who screened positive for a high risk of any sleep disorder were notified by letter as to their risk and provided with contact information for a partnering sleep clinic if they chose to follow-up.
  Arms: Intervention

SUMMARY:
Firefighters work some of the most demanding schedules known under highly stressful and demanding conditions. The need to work frequent extended shifts and long work weeks leads to acute and chronic partial sleep deprivation as well as misalignment of circadian phase. Sleep disorders are common, costly, and treatable, but often remain undiagnosed and untreated and it is likely that a significant proportion of firefighters suffer from undiagnosed sleep disorders which will further impair their sleep and exacerbate fatigue.In the current proposal, we aim to address the health, performance and safety issues related to fatigue in firefighters and test the effectiveness of a Comprehensive Firefighter Fatigue Management Program (CFFMP) that we have termed 'Operation Healthy Sleep.'

DETAILED DESCRIPTION:
We propose to use a station-level, randomized experimental design to test the hypotheses that implementation of a Comprehensive Firefighter Fatigue Management Program will:

1. improve the mean total sleep, alertness and cognitive performance of firefighters;
2. improve firefighter safety, as determined by:

   1. decreased rates of motor vehicle crashes;
   2. decreased on-the-job injuries;
3. improve firefighter performance, as determined by decreased response time;
4. improve firefighters' health, as determined by:

   1. diagnosis and treatment of sleep disorders
   2. improved general health indices
   3. decreased number of 'sick' days
5. improve firefighters' and families' job satisfaction and ability to cope with extended work hours.

ELIGIBILITY:
Inclusion Criteria:

* This proposal includes research involving human subjects (fire department employees).
* Active firefighters working in the study fire department will be eligible to participate in the study.
* All applicants will be considered without bias, regardless of race, ethnicity, or national origin.

Exclusion Criteria:

* Non fire department employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1189 (Actual)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lockley, Ph.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- BWH Division of Sleep Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We invited 73 departments to consider participating based on size and workload, and received 32 responses. Based on interview, selection was based on department cooperation, the practicalities of initiating the program, and the availability of departmental measures for analysis. We selected a mid-sized fire department with ~1200 firefighters.
Pre-assignment Details: 32 fire department stations were paired according to the previous calendar years' workload. One station from each pair (16 stations) was randomly assigned to receive the program. All personnel from the intervention stations were instructed to attend scheduled education sessions.
Groups:
- Intervention: Workplace-based fatigue risk management program consisting of sleep health education and sleep disorders screening.
  32 stations were paired according to workload. One from each pair was randomized to receive the intervention program. Firefighters were instructed to attend an education presentation which provided information on firefighter mortality, fatigue-related hazards and discussed the importance of sleep, and included strategies to improve sleep hygiene and how to use caffeine and naps effectively to promote alertness. Firefighters were then invited to complete a voluntary sleep disorders screening survey. This survey used validated, self-report screening tools for obstructive sleep apnea, moderate to severe insomnia, restless legs syndrome and shift work disorder. All of those who screened positive for a high risk of any sleep disorder were notified by letter as to their risk and provided with contact information for a partnering sleep clinic if they chose to follow-up.
- Control: Current practice.
  Current practice. Firefighters in the Control Stations continued their normal role and were not invited to attend the sleep education and sleep disorders screening program. There was no formal contact with the control group.
  As part of normal operational requirements, a small number of firefighters are reassigned to other stations each day and therefore 18/588 firefighters from control stations happened to be reassigned to an intervention station on the day of the education session and attended the session.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 601 (Intervention participant data obtained from department. Individuals not enrolled for primary aim.) | 588 (Control participant data obtained from department. Individuals were not enrolled.)
Attended Education Session | 542 | 18
Screened for Sleep Disorders | 416 | 15
Completed 1-year Follow-up Survey | 100 | 4
Completed | 601 | 588
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Workplace-based fatigue risk management program consisting of sleep health education and sleep disorders screening
  Sleep disorders education and screening: Firefighters were instructed to attend an education presentation as operations allowed which provided information on firefighter mortality, fatigue-related health hazards and discussed the importance of sleep, and also included strategies to improve sleep hygiene and how to use caffeine and naps effectively to promote alertness. Firefighters were then invited to complete a voluntary sleep disorders screening survey. This survey used validated, self-report screening tools for obstructive sleep apnea, moderate to severe insomnia, restless legs syndrome and shift work disorder. All of those who screened positive for a high risk of any sleep disorder were notified by letter as to their risk and provided with contact information for a partnering sleep clinic if they chose to follow-up.
- Control: Current practice
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 601 | 588 | 1189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (7.3) | 44.4 (7.4) | 43.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 590 | 583 | 1173
Race/Ethnicity, Customized [Number; unit: participants] — The data reflect the categories collected by the fire department
  participants
    White | 541 | 540 | 1081
    Black | 45 | 40 | 85
    Hispanic | 4 | 2 | 6
    Asian | 1 | 3 | 4
    Native American | 3 | 1 | 4
    Biracial | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Firefighters' Health, as Determined by Number of 'Sick' Days Over 12 Months
Description: We assessed 'sick days' cumulatively over 12 months in two ways from departmental payroll records; the number of 24-hour pay periods coded as 'sick' time per firefighter and the number of 24-hr pay periods coded as injury and disability per firefighter. Fewer sick days is indicative of better health.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days/firefighter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 601 | 588
days/firefighter
  Sick days | 3.1 (4.3) | 3.2 (4.5)
  Disability/Injury days | 1.4 (5.9) | 2.6 (8.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Analysis for 'sick' days; Test type: Superiority or Other; p = 0.66, t-test, 2 sided
Statistical Analysis 2: Comparison: Intervention vs Control; Analysis for 'disability/injury' days; Test type: Superiority or Other; p = 0.033, t-test, 2 sided
Statistical Analysis 3: Comparison: Intervention vs Control; Mixed model analysis was conducted for 'disability/injury' days; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mixed model analysis with nested random effects for possible station-level and station-pairing correlation (3-level hierarchical linear model)

2. Primary Outcome: Firefighter Safety, as Determined by Motor Vehicle Crashes Over 12 Months
Description: Fewer motor vehicle crashes is indicative of better health. We assessed motor vehicle crashes cumulatively over 12 months. Accidents were counted as any incident that resulted in the filing and review of a departmental Fleet Accident Report.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: incidents/firefighter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 601 | 588
incidents/firefighter | 0.11 (0.35) | 0.10 (0.31)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.87, t-test, 2 sided

3. Primary Outcome: Firefighter Safety, as Determined by On-the-job Injuries Over 12 Months
Description: Fewer on-the-job injuries is indicative of better health. We assessed injuries cumulatively over 12 months. Injuries that triggered the filing of an official city government accident report as the result of following normal departmental procedures were included in this study.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: injury report/firefighter
Arm/Group | Intervention | Control
Number analyzed (Participants) | 601 | 588
injury report/firefighter | 0.37 (0.63) | 0.40 (0.63)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority or Other; p = 0.31, t-test, 2 sided; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.60 to 0.98] — The Odds Ratio analyses compared the odds of reporting at least one injury during the study between those who did (n=560) and did not (n=629) attend the education sessions, regardless of station assignment (intervention or control)

4. Secondary Outcome: Change in the Mean Total Sleep Time
Description: A higher total sleep time is indicative of better sleep. The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  The analysis for total sleep time is limited to those individuals in the intervention stations who participated in the program, completed both the study start and 12-month follow-up survey, and had at least 1 week of work scheduled in the 4 weeks prior to each survey.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 62/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: Hours/week
Groups:
- Intervention - Study Start: Workplace-based fatigue risk management program consisting of sleep health education and sleep disorders screening
  Sleep disorders education and screening: Firefighters were instructed to attend an education presentation as operations allowed which provided information on firefighter mortality, fatigue-related health hazards and discussed the importance of sleep, and also included strategies to improve sleep hygiene and how to use caffeine and naps effectively to promote alertness. Firefighters were then invited to complete a voluntary sleep disorders screening survey. This survey used validated, self-report screening tools for obstructive sleep apnea, moderate to severe insomnia, restless legs syndrome and shift work disorder. All of those who screened positive for a high risk of any sleep disorder were notified by letter as to their risk and provided with contact information for a partnering sleep clinic if they chose to follow-up.
- Intervention - Post-study Follow-up: Firefighters who completed the voluntary sleep disorders screening survey at the start of the study were invited to complete a subset of questions at the end of the 12-month study.
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 62 | 62
Hours/week | 44.84 (7.05) | 45.98 (6.48)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Of the 100 participants who completed both the pre- and post-study survey (see Patient Flow), only 62 completed answered the question about sleep duration at both time points; Test type: Superiority or Other; p = 0.22, Paired t-test

5. Secondary Outcome: Change in the Mean Alertness and Cognitive Performance of Firefighters - Sleepy During Meetings
Description: A lower number of times reported falling asleep during meetings is indicative of better alertness and cognitive performance.
  The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  The analysis for the number of times individuals reported sleeping during meetings is limited to those individuals in the intervention stations who participated in the program, completed both the study start and 12-month follow-up survey.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 27/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: Incidents/month
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 27 | 27
Incidents/month | 0.41 (1.39) | 0.30 (0.78)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Test type: Superiority or Other; p = 0.65, paired t-test

6. Secondary Outcome: Change in the Mean Alertness and Cognitive Performance of Firefighters - Sleeping on the Telephone
Description: A lower number of times reported sleeping on the telephone is indicative of better alertness and cognitive performance.
  The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  The analysis for the number of times individuals reported sleeping on the telephone is limited to those individuals in the intervention stations who participated in the program, completed both the study start and 12-month follow-up survey.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 88/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: Incidents/month
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 88 | 88
Incidents/month | 0.06 (0.38) | 0.05 (0.26)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Test type: Superiority or Other; p = 0.71, paired t-test

7. Primary Outcome: Firefighters' Performance, as Determined by Response Time Over 12 Months
Description: A lower response time is indicative of better performance.
  Following detailed review of departmental procedures and records, we determined that 'turn-out time' was already very rapid and not considered an accurate measure of firefighters' performance by the department. Similarly, 'clearance time' (time from the start until the end of the event), which could last for many hours, was also not considered an appropriate measure of firefighter' performance in relation to sleep and alertness given the multiple factors, many of which are not under the control of the firefighters, that could affect clearance times. We therefore did not address this aim.
Time Frame: 12 months
Population: Following review of departmental records, we determined that 'turn-out time' and 'clearance time' were not appropriate measures of firefighter' performance in relation to sleep and alertness given the multiple factors that could affect them. We therefore did not address this aim.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Sleep Disorders According to Voluntary Sleep Disorders Screening Questionnaire
Description: Firefighters were instructed to attend a mandatory 30-min education training presentation as operations allowed. Following the education, firefighters were invited and encouraged to complete a voluntary sleep disorders screening questionnaire. This questionnaire used validated, self-report screening tools for Obstructive Sleep Apnea (OSA), moderate to severe insomnia, restless legs syndrome and shift work disorder. All of the respondents who screened positive for a high risk of any sleep disorder were notified by letter as to their risk and provided with contact information for a local American Academy of Sleep Medicine-certified, partnering sleep clinics if they chose to follow-up. Participants were also free to seek medical follow-up elsewhere. Telephone calls were made to all high risk participants to ensure that they were aware of the results, and to facilitate clinic scheduling. Participants were asked to provide voluntary medical records release consent for tracking diagnoses.
Time Frame: Baseline (Study start)
Population: A total of 431 firefighters completed the sleep disorders screening survey including 416 from the intervention stations and 15 who were temporarily assigned to duty in the intervention stations on the day of the survey. We did not consider these 15 firefighters as a separate population.
Measure: Number; unit: participants
Groups:
- Baseline (Intervention): Firefighters in the intervention group who volunteered to complete the sleep disorders screening survey
Arm/Group | Baseline (Intervention)
Number analyzed (Participants) | 431
participants
  Any sleep disorder | 179
  Obstructive Sleep Apnea | 135
  Insomnia | 33
  Restless Legs Syndrome | 15
  Shiftwork Disorder | 40
Statistical Analysis 1: Comparison: Baseline (Intervention); This analysis describes the prevalence of the risk of any sleep disorders; there is no comparison group; Test type: Superiority or Other; Percentage of firefighters screened = 41.5
Statistical Analysis 2: Comparison: Baseline (Intervention); This analysis describes the prevalence of the risk of obstructive sleep apnea only; there is no comparison group; Test type: Superiority or Other; Percentage of firefighters screene = 31.3
Statistical Analysis 3: Comparison: Baseline (Intervention); This analysis describes the prevalence of the risk of insomnia; there is no comparison group; Test type: Superiority or Other; Percentage of firefighters screene = 7.7
Statistical Analysis 4: Comparison: Baseline (Intervention); This analysis describes the prevalence of the risk of restless legs syndrome only; there is no comparison group; Test type: Superiority or Other; Percentage of firefighters screene = 3.5
Statistical Analysis 5: Comparison: Baseline (Intervention); This analysis describes the prevalence of the risk of shiftwork disorder only; there is no comparison group; Test type: Superiority or Other; Percentage of firefighters screene = 9.3

9. Secondary Outcome: Change in the Mean Alertness and Cognitive Performance of Firefighters - Sleeping While Driving
Description: A lower number of times reported sleeping while driving is indicative of better alertness and cognitive performance.
  The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  The analysis for the number of times individuals reported being sleepy while driving is limited to those individuals in the intervention stations who participated in the program, completed both the study start and 12-month follow-up survey.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 81/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: Incidents/month
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 81 | 81
Incidents/month | 0.22 (0.63) | 0.14 (0.65)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Test type: Superiority or Other; p = 0.31, paired t-test

10. Secondary Outcome: Change in the Mean Alertness and Cognitive Performance of Firefighters - Sleeping While Stopped in Traffic
Description: A lower number of times reported sleeping while stopped in traffic is indicative of better alertness and cognitive performance.
  The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  The analysis for the number of times individuals reported sleeping while stopped in traffic is limited to those individuals in the intervention stations who participated in the program, completed both the study start and 12-month follow-up survey.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 82/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: Incidents/month
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 82 | 82
Incidents/month | 0.21 (0.72) | 0.09 (0.36)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Sleeping while stopped in traffic; Test type: Superiority or Other; p = 0.16, Paired t-test, 2-sided

11. Secondary Outcome: Change in Firefighters' Health, as Determined by General Health Indices;
Description: The outcome measure was assessed in the intervention group only at the start and end of the program. There are no data for the control group and therefore they have not been added or reported as a separate study arm.
  A higher health index is indicative of better health. We assessed general health with the question ' In general, would you say your health is Excellent/Very good/Good/Fair/Poor?' and coded the answers from 5-1, respectively.
Time Frame: Baseline to 12 months
Population: Within-subject pre- versus post-study. Only 97/100 individuals in the intervention group who completed the end-of-year survey responded to this question at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 97 | 97
units on a scale | 3.73 (0.82) | 3.68 (0.81)
Statistical Analysis 1: Comparison: Intervention - Study Start vs Intervention - Post-study Follow-up; Test type: Superiority or Other; p = 0.46, Paired t-test, 2-sided

12. Secondary Outcome: Change Firefighters' and Families' Job Satisfaction and Ability to Cope With Extended Work Hours
Description: In developing the study detail with the department, it became apparent that it would be impractical to assess firefighters' and families' job satisfaction and ability to cope with extended work hours in a meaningful way. We therefore did not address this aim.
Time Frame: Baseline to 12 months
Population: In developing the study detail with the department, it became apparent that it would be impractical to assess firefighters' and families' job satisfaction and ability to cope with extended work hours in a meaningful way. We therefore did not address this aim.
Arm/Group | Intervention - Study Start | Intervention - Post-study Follow-up
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Description: A total of 431 firefighters completed the sleep disorders screening survey including 416 from the intervention stations and 15 who were temporarily assigned to duty in the intervention stations on the day of the survey. There was 0 adverse events in either group.
Groups:
- Intervention: Workplace-based fatigue risk management program consisting of sleep health education and sleep disorders screening
  Sleep disorders education and screening: Firefighters were instructed to attend an education presentation which provided information on firefighter mortality, fatigue-related health hazards and discussed the importance of sleep, including strategies to improve sleep hygiene and how to use caffeine and naps effectively to promote alertness. Firefighters were then invited to complete a voluntary sleep disorders screening survey which used validated, self-report screening tools for obstructive sleep apnea, moderate to severe insomnia, restless legs syndrome and shift work disorder. Those who screened positive for any sleep disorder were notified as to their risk and provided with contact information for a partnering sleep clinic if they chose to follow-up. Of the 431 firefighters completed the sleep disorders screening survey, 416 were from the intervention stations.
- Control: A total of 15/588 firefighters in the control stations who were temporarily assigned to duty in the intervention stations on the day of the survey completed the screening survey. The remaining 573 firefighters did not complete the survey and therefore there are no adverse event data to report.
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/416 | 0/15
Other Adverse Events (participants affected / at risk) | 0/416 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No